CLINICAL TRIAL: NCT04045548
Title: Benefits of Vaginal Dinoprostone Administration Prior to Levonorgestrel-releasing Intrauterine System Insertion in Women Delivered Only by Elective Cesarean Section: a Randomized Double-blind Clinical Trial.
Brief Title: Vaginal Dinoprostone Administration Prior to Insertion Levonorgestrel-releasing Intrauterine System in Women With no Previous Vaginal Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone IUD
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Intrauterine Device
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 2 hours before IUD insertion.
  Interventions: Drug: Dinoprostone
- placebo (Placebo Comparator): one tablet of placebo inserted by the study nurse 2 hours before IUD insertion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dinoprostone — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 6 hours before IUD insertion.
  Arms: dinoprostone
Drug: Placebo — one tablet of placebo inserted by the study nurse 6 hours before IUD insertion.
  Arms: placebo

SUMMARY:
To investigate whether vaginal dinoprostone administered before the levonorgestrel-releasing intrauterine system(IUs) insertion reduces failed insertions, insertion-related complications, and pain in Women With no Previous Vaginal Delivery.

DETAILED DESCRIPTION:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women
* Women that did not receive any analgesics or Dinoprostone in the 24 hours prior to insertion
* Women who delivered only by cesarean section

Exclusion Criteria:

* Women with any uterine abnormalities as congenital anomalies, endometrial lesions, adenomyosis, fibroids.
* Those with a Category 3 or 4 conditions for intrauterine device insertion according to the WHO Medical Eligibility Criteria for contraceptive use
* Allergy to dinoprostone.
* Women refuse to participate in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores during intrauterine device insertion | 10 minutes
  The difference in pain scores during intrauterine device insertion using visual analog scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Cairo, Egypt